CLINICAL TRIAL: NCT03131635
Title: Effectiveness of a Developmental Reciprocity Treatment Program in Autism
Acronym: DRTP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated (halted prematurely) due to COVID-19.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Antonio Hardan, Professor of Psychiatry and Behavioral Sciences, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 40026
Record Dates: First submitted 2017-04-24; First posted 2017-04-27 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Autism Spectrum Disorder; Autism
Keywords: Developmental
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Developmental Reciprocity Treatment Program (DRT-P) (Experimental): Developmental Reciprocity Treatment is an early intervention that applies developmentally-informed teaching methods in naturalistic settings in order to target social and communication deficits.
  Interventions: Behavioral: Developmental Reciprocity Treatment Program (DRT-P)
- Delayed Treatment Group (DTG) (No Intervention)

INTERVENTIONS:
Behavioral: Developmental Reciprocity Treatment Program (DRT-P) — Developmental Reciprocity Treatment is an early intervention that applies developmentally-informed teaching methods in naturalistic settings in order to target social and communication deficits.
  Arms: Developmental Reciprocity Treatment Program (DRT-P)

SUMMARY:
This is a research study examining the effectiveness of a Developmental Reciprocity Treatment Program (DRT-P) in treating social deficits in children with Autism Spectrum Disorders (ASD). Developmental Reciprocity Treatment is an early intervention that applies developmentally-informed teaching methods in naturalistic settings in order to target social and communication deficits.

Researchers have begun to develop strategies to investigate the effectiveness of combining a parent training program teaching parents how to implement DRP with in-home, therapist-implemented treatment. To determine the effectiveness of the DRT-P, it will be compared to a delayed treatment group (DTG) by conducting a randomized controlled 24-week trial. This research will allow us to help in the development of therapeutic approaches that can meet the increasing service demands for families. We hope that investigating interventions that aim to improve core deficits will aid in providing better care for children with autism.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Autism Spectrum Disorder based on Autism Diagnostic Interview Revised (ADI-R), Autism Diagnostic Observation Schedule (ADOS-2), DSM-5, and expert clinical opinion;
* Males and females in good medical health between 2.0 and 5 years 11 months;
* Ability to participate in the testing procedures to the extent that valid standard scores can be obtained;
* Stable treatment (e.g., applied behavior analysis), speech therapy, psychotropic medication(s) or biomedical intervention(s) for at least 1 month prior to baseline measurements with no anticipated changes during study participation;
* Availability of at least one English-speaking parent who can consistently participate in parent training and research measures;
* Clinical Global Impression(CGI) Severity Social Interaction and Communication Integrated Subscale ≥4;
* Meet the cutoff for Autism on the ADOS-2.

Exclusion Criteria:

* Current or lifetime diagnosis of severe psychiatric disorder (e.g., bipolar disorder, etc.);
* A well-established genetic syndrome, such as Fragile X;
* Presence of active medical problem (e.g., unstable seizure disorder or heart disease);
* Child's primary language other than English;
* Previous adequate trial or training of a developmentally based intervention;
* Participants living more than 45 miles from Stanford University;
* Children with more than 20 hours of in-home ABA;
* At least one room of the house must be available to be dedicated to treatment during session times;
* There must be no serious health and safety risks present in the home environment;
* The research team has the right to refuse to perform sessions in-home even if the criteria above are met.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2020-07-16 (Actual); Study Completion 2020-07-16 (Actual)

PRIMARY OUTCOMES:
Change from Baseline on the Social Responsiveness Scale (SRS) at 6, 12, and 24 weeks | Baseline, 6, 12, and 24 weeks
Change from Baseline on the Brief Observation of Social Communication Change (BOSCC) at 24 weeks | Baseline and 24 weeks

SECONDARY OUTCOMES:
Change from Baseline on the Vineland Adaptive Behavior Scales, Second Edition (VABS-II) at 12, and 24 weeks | Baseline, 12, and 24 weeks
Change from Baseline on the Stanford Social Dimensions Scale (SSDS) Questionnaire. | Baseline, 12, and 24 weeks

OTHER OUTCOMES:
Change from Baseline on the Structured Lab Observation (SLO) at 6, 12, and 24 weeks | Baseline, 6, 12, and 24 weeks
Change from Baseline on the Mullen Scales of Early Learning at 24 weeks | Baseline and 24 weeks
Change from Baseline on the MacArthur-Bates Communication Development Inventory at 12, and 24 weeks | Baseline, 12, and 24 weeks
Change from Baseline on the Behavior Rating Inventory of Executive Function, Preschool (BRIEF-P) at 12, and 24 weeks | Baseline, 12, and 24 weeks
Change from Baseline on the Clinical Global Impression Scale at 12, and 24 weeks | Baseline, 12, and 24 weeks
Change from Baseline on the Family Empowerment Scale (FES) at 12, and 24 weeks | Baseline, 12, and 24 weeks
Change from Baseline on the Social attention and word-learning eye tracking task at 12, and 24 weeks | Baseline, 12, and 24 weeks
Change from Baseline on the Short Sensory Profile Questionnaire (SSPQ) at 12, and 24 weeks | Baseline, 12, and 24 weeks
Change from Baseline on the Parenting Stress Index (PSI) at 12, and 24 weeks | Baseline, 12, and 24 weeks
Change from Baseline on the Aberrant Behavior Checklist (ABC) at 12, and 24 weeks | Baseline, 12, and 24 weeks
Change from Baseline on the Repetitive Behavior Scale Revised (RBS-R) at 12, and 24 weeks | Baseline, 12, and 24 weeks
Change from Baseline on the Pediatric Quality of Life Scale at 12, and 24 weeks | Baseline, 12, and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Y. Hardan, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No